CLINICAL TRIAL: NCT00131664
Title: Avandia™ + Amaryl™ or Avandamet™ Compared With Metformin: A 48-week Randomized, Open-label, Multicentre Phase IIIB Study to Compare the Effectiveness of Combination Therapy to Monotherapy in Type 2 Diabetes Mellitus Patients
Brief Title: Avandia™ + Amaryl™ or Avandamet™ Compared With Metformin (AVALANCHE™ Study)
Acronym: AVALANCHE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Heart Research Centre (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Dr. Anatoly Langer, Chair, Steering Committe, Canadian Heart Research Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVM103436
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Results first posted 2013-04-17 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rosiglitazone-metformin combination; Rosiglitazone; Metformin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Avandamet (Active Comparator): Avandamet 2 mg / 500 mg twice daily titration up to 4 mg / 1000 mg twice daily over 6 months
  Interventions: Drug: Avandamet
- Avandia and Amaryl (Active Comparator): Avandia + Amaryl 4 mg + 1 mg once daily titration up to 8 mg + 2 mg once daily over 6 months
  Interventions: Drug: Avandia and Amaryl
- Metformin (Active Comparator): Metformin 500 mg twice daily titration up to 1000 mg twice daily over 6 months
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Avandamet — Avandamet 2 / 500 mg twice daily titration up to 4 mg / 1000 mg twice daily compared to Avandia 4 mg and Amaryl 1 mg once daily over 6 months or compared to Metformin 500 mg twice daily up to 1000 mg over 6 months.
  Other Names: rosiglitazone maleate and metformin hydrochloride; Avandamet 2 mg / 500 mg; Avandamet 4 mg / 500 mg; Avandamet 4 mg / 1000 mg
  Arms: Avandamet
Drug: Avandia and Amaryl — Avandia 4 mg and Amaryl 1 mg once daily compared to Avandamet 2 / 500 mg twice daily titration up to 4 mg / 1000 mg twice daily, or compared to Metformin 500 mg twice daily up to 1000 mg over 6 months.
  Other Names: rosiglitazone maleate and glimepiride; Avandia (rosiglitazone maleate) 4 mg; Avandia (rosiglitazone maleate) 8 mg; Amaryl (glimepiride) 1 mg; Amaryl (glimepiride) 2 mg; Amaryl (glimepiride) 4 mg
  Arms: Avandia and Amaryl
Drug: Metformin — Metformin 500 mg twice daily up to 1000 mg over 6 months compared to Avandia 4 mg and Amaryl 1 mg once daily or compared to Avandamet 2 / 500 mg twice daily titration up to 4 mg / 1000 mg twice daily
  Other Names: Metformin 500 mg; Metformin 850 mg
  Arms: Metformin

SUMMARY:
The incidence of type 2 diabetes is on the increase. According to recent Canadian Diabetes Association guidelines glucose control, based on the A1C measurement, needs to be achieved within a 6-12 month period of time after the initial diagnosis of type 2 diabetes. The guidelines on the use of antihyperglycemic agents identify the potential benefits of sub-maximal oral combination therapy in order to achieve more rapid and improved glycemic control compared with higher dose monotherapy. Furthermore, many patients on prolonged oral antihyperglycemic monotherapy who then start on combination therapy may not achieve the required target glycemic control. Indeed early initiation of combination therapies may be necessary to achieve and maintain glycemic targets because of the progressive deterioration of pancreatic β cell function and glycemic control.

DETAILED DESCRIPTION:
AvandametTM combines two oral antihyperglycemic agents, rosiglitazone maleate and metformin hydrochloride, with different but complementary mechanisms of action to improve glycemic control while reducing circulating insulin levels in patients with type 2 diabetes. AvandiaTM and AmarylTM combine two antidiabetic agents, rosiglitazone maleate and glimepiride. Glimepiride is an effective antihyperglycemic agent which has a low incidence of hypoglycemia, symptomatic hypoglycemia, severe hypoglycemia, and confirmed hypoglycemia. Subjects in this study who are inadequately controlled on diet, exercise and a submaximal dose of metformin or sulfonylurea (SU) will be randomized to either a combination of metformin plus rosiglitazone (AvandametTM) or a combination of AvandiaTM + AmarylTM or a Metformin monotherapy arm. As per the Canadian Diabetes Association (CDA) guidelines, their fasting plasma glucose and A1C to be 7 (mmol/L / percent) or less throughout the study. If the subject does not achieve the target then either AvandametTM or AvandiaTM and AmarylTM or Metformin will be up-titrated in an effort to reach this CDA recommended target. This study will attempt to demonstrate that the either combination arm of rosiglitazone plus metformin (AvandametTM) or the other combination arm of AvandiaTM + AmarylTM will provide greater glycemic control while avoiding the side-effects associated with the use of maximal dose metformin.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes patients
2. 18 - 75 years old
3. Type 2 diabetes mellitus (DM) drug naïve or on submaximal oral monotherapy < 3 years
4. A1C criteria at screening:

   1. 7.1-10% for drug naïve patients after failure of diet control and life-style modification
   2. 7.1 - 9% on single therapy (e.g. not more 10 mg of Glyburide or 4 mg of Amaryl™ or 1000mg of Metformin) who will start after 2 weeks wash-out. During wash out the following will be done: i) diet and life style modification ii) Angiotensin converting enzyme inhibitor (ACE), aspirin (80 mg), and statin if appropriate
5. Signed informed consent

Exclusion Criteria:

1. Type 1 diabetes
2. Subjects currently treated with insulin
3. Subject treated for previous 3 month with any thiazolidinedione (TZD)
4. Evidence of clinically significant concomitant illnesses which are not controlled by medication and/or may limit participation in the study as judged by the investigator
5. Subjects who have hypersensitivity to any components of study drugs
6. Participation in a clinical trial and/or intake of an investigational drug within 30 days prior to screening.
7. Pregnant or nursing females
8. Females of childbearing potential who are not on adequate birth control
9. Liver enzymes (Alanine Aminotransferase (ALT) > 2.5 times upper limit of normal)
10. Renal impairment: serum creatinine ≥ 136umol/L (males) and ≥ 124 umol/L (females)
11. Congestive Heart Failure (CHF class III/IV)
12. Weight >160 kg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2005-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: robert josse, md, Principal Investigator — University of Toronto
Locations (1):
- Canadian Heart Research Centre, Toronto, Ontario, Canada

REFERENCES:
- See also: coordinating centre web site — http://www.chrc.net

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 391 patients were randomized from 49 Canadian sites of General Practitioners and Community Endocrinologists during an 8 month recruitment period.
Pre-assignment Details: This open-label, prospective, randomized multi-centre study included naïve or recently treated type 2 diabetes mellitus (T2DM) patients. Recently treated patients (up to 3 years on single therapy of a low to moderate dose of Glyburide or Amaryl™ or Metformin) entered the study after a 2-week wash-out period.
Groups:
- Avandia and Amaryl: Avandia™ + Amaryl™ Arm: at month 2 initial dose of 4 mg + 1 mg once daily (OD) was titrated up to 8 mg + 1 mg OD; at month 4 it was further titrated up to 8 mg + 2 mg OD.
- Avandamet: Avandamet™ Arm: at month 2 the initial dose of 2 mg / 500 mg twice daily (BID) was titrated up to 4 mg / 500 mg BID; at month 4 it was be further titrated up to 4 mg / 1000 mg BID.
- Metformin: Metformin Arm: initial dose of 500 mg twice daily (BID) was titrated up to 850 mg BID at month 2. At month 4, it was further titrated up to 1000 mg BID.
- Avandia, Amaryl and Metformin: Avandia™ + Amaryl™ Arm: At month 6, if patients not achieving A1C target of less than 7 received additional specified drug therapy. Metformin was added and titrated up to 1000 mg twice daily (BID) maximum dose for an additional 6 months.
- Avandamet and Amaryl: Avandamet™ Arm: At month 6, if patients not achieving A1C target of less than 7 received additional specified drug therapy. Amaryl™ was added and titrated up to 4 mg once daily maximum dose for an additional 6 months
- Metformin and Amaryl: Metformin Arm: At month 6, if patients not achieving A1C target of less than 7 received additional specified drug therapy. Amaryl™ was added and titrated up to 4 mg once daily maximum dose for an additional 6 months.
Period: First Period (First 6 Months)
Arm/Group | Avandia and Amaryl | Avandamet | Metformin | Avandia, Amaryl and Metformin | Avandamet and Amaryl | Metformin and Amaryl
Started | 136 | 135 | 120 | 0 | 0 | 0
Completed | 111 | 117 | 104 | 0 | 0 | 0
Not Completed | 25 | 18 | 16 | 0 | 0 | 0
Not completed — Lost to Follow-up | 7 | 3 | 3 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 2 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 6 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 9 | 4 | 5 | 0 | 0 | 0
Not completed — Clinically significant lab abnormalities | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Administrative reasons | 2 | 0 | 5 | 0 | 0 | 0
Period: Second Period (Additional Drug Added)
Arm/Group | Avandia and Amaryl | Avandamet | Metformin | Avandia, Amaryl and Metformin | Avandamet and Amaryl | Metformin and Amaryl
Started | 90 (21 had added Metformin at Month 6) | 101 (16 had added Amaryl at Month 6) | 79 (25 had added Amaryl at Month 6) | 21 | 16 | 25
Completed | 81 | 97 | 76 | 19 | 15 | 22
Not Completed | 9 | 4 | 3 | 2 | 1 | 3
Not completed — Lost to Follow-up | 3 | 0 | 2 | 1 | 0 | 2
Not completed — Protocol Violation | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Clinically significant lab abnormalities | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Administrative reasons | 4 | 2 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Avandia and Amaryl: 4 mg + 1 mg once daily titration up to 8 mg + 2 mg once daily over 6 months
- Avandamet: 2 mg / 500 mg twice daily titration up to 4 mg / 1000 mg twice daily over 6 months
- Metformin: 500 mg twice daily titration up to 1000 mg twice daily over 6 months
- Total: Total of all reporting groups
Arm/Group | Avandia and Amaryl | Avandamet | Metformin | Total
Number analyzed (Participants) | 136 | 135 | 120 | 391
Age Continuous [Mean (Standard Deviation); unit: years] | 54.3 (10.1) | 53.7 (11.6) | 56.0 (10.1) | 54.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 59 | 57 | 164
  Male | 88 | 76 | 63 | 227
Region of Enrollment [Number; unit: participants]
  Canada | 136 | 135 | 120 | 391

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in A1C at Month 6
Description: Change from baseline was calculated as the Month 6 value minus the baseline value, with last on-treatment observation carried forward (LOCF) from Month 2 for withdrawn subjects or missing values.
Time Frame: Baseline and Month 6
Population: Intent-to-Treat (ITT) population: all randomized subjects who took at least one dose of study medication and had at least one valid observation. For withdrawn subjects or missing values, the last on-treatment observation was carried forward (LOCF). Only subjects with a value at baseline and at Month 6 were analyzed.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Number analyzed (Participants) | 125 | 128 | 115
percent
  Baseline | 8.14 (0.095) | 7.96 (0.076) | 7.90 (0.085)
  Change from baseline | -1.61 (0.108) | -1.39 (0.081) | -1.02 (0.092)

2. Secondary Outcome: Mean Change From Baseline in A1C at Month 4
Description: Change from baseline was calculated as the Month 4 value minus the baseline value, with last on-treatment observation carried forward (LOCF) from Month 2 for withdrawn subjects or missing values.
Time Frame: Baseline and Month 4
Population: Intent-to-Treat (ITT) population: all randomized subjects who took at least one dose of study medication and had at least one valid observation. For withdrawn subjects or missing values, the last on-treatment observation was carried forward (LOCF). Only subjects with values at baseline and Month 4 were analyzed.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Number analyzed (Participants) | 125 | 128 | 115
percent | -1.44 (0.099) | -1.28 (0.083) | -0.94 (0.097)

3. Secondary Outcome: Mean Change From Baseline in A1C at Month 12
Description: Change from baseline was calculated as the Month 12 value minus the baseline value, with last on-treatment observation carried forward (LOCF) from Month 2 for withdrawn subjects or missing values.
Time Frame: Baseline and Month 12
Population: Intent-to-Treat (ITT) population: all randomized subjects who took at least one dose of study medication and had at least one valid observation. For withdrawn subjects or missing values, the last on-treatment observation was carried forward (LOCF). Only subjects with values at baseline and Month 12 were analyzed.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Number analyzed (Participants) | 131 | 131 | 116
percent | -1.50 (0.115) | -1.56 (0.086) | -1.14 (0.111)

4. Secondary Outcome: Number of Subjects Achieving A1C Target at Month 4
Description: A1C responders were described as subjects having achieved A1C less than 7 percent at Month 4, with LOCF from Month 2.
Time Frame: Month 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Number analyzed (Participants) | 125 | 128 | 115
participants | 83 | 96 | 69

5. Secondary Outcome: Number of Subjects Achieving A1C Target at Month 6
Description: A1C responders were described as subjects having achieved A1C less than 7 percent at Month 6, with LOCF from Month 2.
Time Frame: Month 6
Population: Intent-to-Treat (ITT) population: all randomized subjects who took at least one dose of study medication and had at least one valid observation. For withdrawn subjects or missing values, the last on-treatment observation was carried forward (LOCF). Only subjects with values at baseline Month 6 were analyzed.
Measure: Number; unit: participants
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Number analyzed (Participants) | 125 | 128 | 115
participants | 94 | 98 | 69

6. Secondary Outcome: Number of Subjects Achieving A1C Target at Month 12
Description: A1C responders were described as subjects having achieved A1C less than 7 percent at Month 12 with LOCF from Month 2.
Time Frame: Month 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Number analyzed (Participants) | 131 | 131 | 116
participants | 95 | 111 | 82

7. Secondary Outcome: Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Month 4
Description: as for outcome 2
Time Frame: Baseline and Month 4
Population: as for outcome 2
Measure: Mean (Standard Error); unit: millimoles per litre (mmol/L)
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Number analyzed (Participants) | 124 | 127 | 115
millimoles per litre (mmol/L) | -2.86 (0.247) | -2.33 (0.181) | -1.75 (0.204)

8. Secondary Outcome: Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Month 6
Description: as for outcome 1
Time Frame: Baseline and Month 6
Population: Intent-to-Treat (ITT) population: all randomized subjects who took at least one dose of study medication and had at least one valid observation. For withdrawn subjects or missing values, the last on-treatment observation was carried forward (LOCF). Only subjects with values at baseline and Month 6 were analyzed.
Measure: Mean (Standard Error); unit: millimoles per litre (mmol/L)
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Number analyzed (Participants) | 124 | 127 | 115
millimoles per litre (mmol/L) | -2.98 (0.259) | -2.55 (0.200) | -1.86 (0.192)

9. Secondary Outcome: Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Month 12
Description: Change from baseline was calculated as the Month 12 value minus the baseline value, with LOCF from Month 2 for withdrawn subjects or missing values.
Time Frame: Baseline and Month 12
Population: as for outcome 8
Measure: Mean (Standard Error); unit: millimoles per litre (mmol/L)
Groups:
- Avandia and Amaryl: 2 mg / 500 mg twice daily titration up to 4 mg / 1000 mg twice daily over 6 months
- Avandamet: 4 mg + 1 mg once daily titration up to 8 mg + 2 mg once daily over 6 months
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Number analyzed (Participants) | 130 | 130 | 116
millimoles per litre (mmol/L) | -2.71 (0.274) | -2.76 (0.225) | -2.12 (0.231)

10. Secondary Outcome: Number of Subjects Achieving FPG Target at Month 4
Description: FPG responders were described as subjects having achieved FPG less than 7 mmol/L at Month 4 with LOCF from Month 2.
Time Frame: Month 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Number analyzed (Participants) | 124 | 127 | 115
participants | 58 | 65 | 38

11. Secondary Outcome: Number of Subjects Achieving FPG Target at Month 6
Description: FPG responders were described as subjects having achieved FPG less than 7 mmol/L at Month 6 with LOCF from Month 2.
Time Frame: Month 6
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Number analyzed (Participants) | 124 | 127 | 115
participants | 61 | 76 | 43

12. Secondary Outcome: Number of Subjects Achieving FPG Target at Month 12
Description: FPG responders were described as subjects having achieved FPG less than 7 mmol/L at Month 12 with LOCF from Month 2.
Time Frame: Month 12
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Number analyzed (Participants) | 130 | 130 | 116
participants | 64 | 86 | 51

13. Secondary Outcome: Mean Change From Baseline in 5 Year UKPDS Risk Scores at Month 6
Description: Change from baseline was calculated as the Month 6 value minus the baseline value, with LOCF from Month 2. The UKPDS (United Kingdom Prospective Diabetes Study) risk engine calculated was based on 5 years risk using gender, race, age at diagnosis of diabetes, duration of diabetes, smoking status, A1C, systolic blood pressure and total cholesterol to high-density lipoprotein (HDL) ratio at a specified visit.
  The UKPDS cardiovascular disease (CVD) risk engine is used to estimate the risk of having coronary heart disease in type II diabetes according to the UKPDS model. The possible risk scores can range from 0 to 100% and hence lower scores would predict a person is less likely to have an event.
Time Frame: Baseline and Month 6
Population: as for outcome 8
Measure: Mean (Standard Error); unit: percent
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Number analyzed (Participants) | 111 | 116 | 99
percent | -1.09 (0.246) | -1.05 (0.169) | -1.54 (0.234)

14. Secondary Outcome: Mean Change From Baseline in 5 Year UKPDS Risk Scores at Month 12
Description: Change from baseline was calculated as the Month 12 value minus the baseline value, with LOCF from Month 2. The UKPDS (U.K. Prospective Diabetes Study) risk engine calculated was based on 5 years risk using gender, race, age at diagnosis of diabetes, duration of diabetes, smoking status, A1C, systolic blood pressure and total cholesterol to HDL ratio at a specified visit.
  The UKPDS cardiovascular disease (CVD) risk engine is used to estimate the risk of having coronary heart disease in type II diabetes according to the UKPDS model. The possible risk scores can range from 0 to 100% and hence lower scores would predict a person is less likely to have an event.
Time Frame: Baseline and Month 12
Population: as for outcome 3
Measure: Mean (Standard Error); unit: percent
Groups:
- Metformin: : 500 mg twice daily titration up to 1000 mg twice daily over 6 months
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Number analyzed (Participants) | 122 | 124 | 104
percent | -0.72 (0.392) | -0.62 (0.252) | -1.11 (0.234)

15. Secondary Outcome: Mean Change From Baseline in C-reactive Protein (CRP) at Month 6
Description: Change from baseline was calculated as the Month 6 value minus the baseline value. LOCF was not used for this analysis. CRP was only done at baseline, months 6 and 8. The test was optional and performed only by participating sites.
Time Frame: Baseline and Month 6
Population: All Primary and secondary endpoints were calculated on the Intent to Treat (ITT) population where each patient had at least one dose of the medication and at least one valid observation. Missing values were carried forward (using Last Observation Carried Forward method) except for the calculation of the composite variables.
Measure: Mean (Standard Error); unit: milligram per decilitre (mg/dL)
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Number analyzed (Participants) | 24 | 28 | 22
milligram per decilitre (mg/dL) | -1.20 (0.419) | -1.68 (0.640) | -1.25 (0.804)

16. Secondary Outcome: Mean Change From Baseline in C-reactive Protein (CRP) at Month 12
Description: Change from baseline was calculated as the Month 12 value minus the baseline value, with LOCF from Month 6. CRP was only done at baseline, months 6 and 12. The test was optional and performed only by participating sites.
Time Frame: Baseline and Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Number analyzed (Participants) | 32 | 30 | 25
mg/dL | -0.40 (0.323) | -1.52 (0.642) | -1.52 (0.817)

17. Secondary Outcome: Mean Change From Baseline in Adiponectin at Month 6
Description: Change from baseline was calculated as the Month 6 value minus the baseline value. LOCF was not used for this analysis. Adiponectin was only done at baseline, months 6 and 12. The test was optional and performed only by participating sites.
Time Frame: Baseline and Month 6
Population: as for outcome 8
Measure: Mean (Standard Error); unit: microgram per millilitre (µg/mL)
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Number analyzed (Participants) | 25 | 23 | 22
microgram per millilitre (µg/mL) | 5.73 (0.869) | 6.37 (1.453) | 0.23 (0.299)

18. Secondary Outcome: Mean Change From Baseline in Adiponectin at Month 12
Description: Change from baseline was calculated as the Month 12 value minus the baseline value, with LOCF from Month 6. Adiponectin was only done at baseline, months 6 and 12. The test was optional and performed only by participating sites.
Time Frame: Baseline and Month 12
Population: as for outcome 3
Measure: Mean (Standard Error); unit: µg/mL
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Number analyzed (Participants) | 31 | 27 | 24
µg/mL | 4.95 (0.902) | 8.21 (1.804) | 1.453 (0.371)

ADVERSE EVENTS:
Groups:
- Avandia and Amaryl: Avandia™ + Amaryl™ Arm: at month 2 initial dose of 4 mg +1 mg OD was titrated up to 8 mg + 1 mg OD; at month 4 it was further titrated up to 8 mg / 2 mg OD. At month 6, patients not achieving target received additional specified drug therapy: Metformin was added and titrated up to 1000 mg BID maximum dose for an additional 6 months.
- Avandamet: Avandamet™ Arm: at month 2 the initial dose of 2 mg / 500 mg BID was titrated up to 4 mg / 500 mg BID; at month 4 it was be further titrated up to 4 mg / 1000 mg BID. At month 6, patients not achieving target received additional specified drug therapy Amaryl™ was added and titrated up to 4 mg OD maximum dose for an additional 6 months
- Metformin: Metformin Arm: initial dose of 500 mg BID was titrated up to 850 mg BID at month 2. At month 4, it was further titrated up to 1000 mg BID. At month 6 (visit 6), patients not achieving target received additional specified drug therapy: Amaryl™ was added and titrated up to 4 mg OD maximum dose for an additional 6 months.
Arm/Group | Avandia and Amaryl | Avandamet | Metformin
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/135 | 0/120
Other Adverse Events (participants affected / at risk) | 2/136 | 3/117 | 0/104
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avandia and Amaryl (N=136) | Avandamet (N=117) | Metformin (N=104)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0) — Fractures were all wrist or ankle.

LIMITATIONS AND CAVEATS:
The LOCF used in the ITT population for withdrawn subjects or missing values was analyzed as per protocol. The 3 treatment groups used throughout the results section were the numbers where the patients were originally randomized to.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No